CLINICAL TRIAL: NCT01465009
Title: Double-blind, Randomized, Placebo-controlled, Single Dose, Parallel Group Study Evaluating Efficacy and Safety of 1000 mg Acetylsalicylic Acid and 1000 mg Paracetamol in Adult Patients With Sore Throat Associated With a Common Cold
Brief Title: Placebo and Active Controlled Study to Compare the Efficacy of Aspirin and Paracetamol in Treatment of Sore Throat Associated With a Common Cold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11381
Record Dates: First submitted 2011-05-17; First posted 2011-11-04 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2011-11

CONDITIONS: Common Cold; Pharyngitis; Tonsillitis
Keywords: Sore Throat
MeSH Terms: conditions — Common Cold; Pharyngitis; Tonsillitis | interventions — Aspirin; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465)
- Arm 2 (Active Comparator)
  Interventions: Drug: Paracetamol
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) — Single Administration of 2 tablets Acetylsalicylic acid (500 mg each); in addition, 2 tablets matching placebo to Paracetamol
  Arms: Arm 1
Drug: Paracetamol — Single Administration of 2 tablets Paracetamol (500 mg each); in addition, 2 tablets matching placebo to Acetylsalicylic Acid
  Arms: Arm 2
Drug: Placebo — Single Administration of 2 tablets matching Placebo to Acetylsalicylic Acid together with 2 tablets matching placebo to Paracetamol
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine the efficacy and safety of 1000 mg Aspirin (study medication) by comparing 1000 mg Paracetamol (study medication) in treating the symptoms of sore throat associated with a common cold. The study is designed to develop a treatment method against sore throat associated with a common cold which will have more advantages for patients than the methods that are currently available.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Onset of common cold within the past 5 days
* Current sore throat
* Confirmed presence of a tonsillo-pharyngitis

Exclusion Criteria:

* Hypersensitivity to acetylsalicylic acid, salicylates, paracetamol, or any other NSAID
* Pregnant or lactating women
* History or acute state of peptic ulceration or gastrointestinal bleeding
* History of bleeding tendency
* History of asthma
* Inability to breathe through the nose or a history of chronic mouth breathing
* Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2003-11; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference to baseline of Acetylsalicylic Acid in comparison to Paracetamol | For 6 hours after drug intake

SECONDARY OUTCOMES:
Pain intensity difference to baseline of Acetylsalicylic Acid in comparison to Placebo | For 6 hours after drug intake
Total pain relief of Acetylsalicylic Acid in comparison to Paracetamol | For 6 hours after drug intake
Total pain relief of Acetylsalicylic Acid in comparison to Placebo | For 6 hours after drug intake
Evaluation of Upper Respiratory Tract Infection symtoms | 2 hours after drug intake
Adverse Event collection | Up to 17 days after Screening

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United Kingdom (7):
  - Reading, Berkshire
  - Manchester, Greater Manchester
  - Chorley, Lancashire
  - Wigan, Lancashire
  - Liverpool, Merseyside
  - Cardiff, South Glamorgan
  - Birmingham, West Midlands